CLINICAL TRIAL: NCT03167788
Title: A RANDOMISED CONTROLLED TRIAL OF RED CELL REJUVENATION FOR THE ATTENUATION OF TRANSFUSION ASSOCIATED ORGAN INJURY IN CARDIAC SURGERY: The REDJUVENATE Trial
Brief Title: Red Cell Rejuvenation for the Attenuation of Transfusion Associated Organ Injury in Cardiac Surgery
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Manufacturing Issues
Sponsor: University of Leicester (Other)
Collaborators: National Health Service, United Kingdom (Other Government); Zimmer Biomet (Industry); British Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 0582
Record Dates: First submitted 2017-05-12; First posted 2017-05-30 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2020-05

CONDITIONS: Organ Failure, Multiple; Inflammation; Sepsis
MeSH Terms: conditions — Multiple Organ Failure; Inflammation; Sepsis | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Cross-matched allogeneic stored red cells will be rejuvenated using rejuvesol® Red Blood Cell Processing Solution (Citra Labs, MA, a Zimmer Biomet Company, IN, USA) with washing and re-suspension in an additive solution prior to transfusion. The rejuvenated red cells will then be administered to the patient as per standard practice and according to established institutional protocols. A maximum of 6 rejuvenated red cell units will be transfused within any 24 hour period.
  Interventions: Device: rejuvesol Solution
- Control (Active Comparator): Standard care i.e. Cross-matched allogeneic stored non-rejuvenated, unwashed red cells will be administered to the patient as per standard practice and according to established institutional protocols.
  Interventions: Other: Standard Care

INTERVENTIONS:
Device: rejuvesol Solution — The rejuvenation process involves incubation of stored red cells with a rejuvenating solution, rejuvesol Red Blood Cell Processing Solution (rejuvesol® Solution), Citra labs, MA, a Zimmer Biomet Company, IN, USA) which restores red cell adenosine triphosphate (ATP), 2,3-DPG (diphosphoglycerate), oxygen transfer characteristics and rheology. Post rejuvenation red cells are washed to remove the rejuvesol Solution, and cells are re-suspended in additive solution for transfusion.
  Arms: Intervention
Other: Standard Care — Allogeneic red cells, harvested in citrate-phosphate-dextrose (CPD), leucocyte depleted, saline-adenine-glucose-mannitol (SAGM) stored red cell units, issued by National Health Service Blood & Transplant (NHSBT) will be administered to cardiac surgery patients as per standard practice, and according to established unit protocols.
  Arms: Control

SUMMARY:
The REDJUVENATE Trial proposes to test the hypothesis that postoperative organ injury and inflammation will be less if patients undergoing cardiac surgery who are at risk of large volume blood transfusion (defined as the administration of ≥4 units of red cells) receive rejuvenated washed cells compared to standard care (unwashed aged stored cells).

DETAILED DESCRIPTION:
In the REDJUVENATE trial, we propose to establish whether the administration of rejuvenated red cells will reduce inflammation and organ injury in cardiac surgery patients at risk of large volume blood transfusion when compared to standard care. Organ injury and sepsis accounts for the majority of all deaths following cardiac surgery. Once organ injury is established care is primarily supportive and there are no effective treatments. Prevention is therefore a key clinical strategy to prevent death, morbidity and high healthcare costs attributable to these complications. Sepsis and inflammatory organ injury are also the principal causes of death following paediatric cardiac surgery, trauma, non-cardiac complex surgical procedures and in critical care; clinical settings that are also among the principal consumers of blood components. National and international blood management strategies are focused on these patients. Evidence of a clinical benefit attributable to the use of rejuvenated red cells in cardiac surgery patients is therefore likely to translate into more widespread benefits to patients and the National Health Service (NHS).

ELIGIBILITY:
Inclusion Criteria:

1. Adult cardiac surgery patients (≥18 years) undergoing cardiac surgery with cardiopulmonary bypass.
2. Identified as representing a high risk group for massive blood transfusion using a modified risk score. A large volume blood transfusion (LVBT) score of >23 indicates predicted risk of receiving ≥4 units of allogeneic red cells equal to or greater than 55 per cent.

Exclusion Criteria:

1. Emergency or salvage procedure
2. Patients with end stage renal failure defined as an estimated Glomerular Filtration rate (eGFR) <15 mL/min/1.72 m2 calculated from the Modification of Diet in Renal Disease equation, or patients who are on long-term haemodialysis or have undergone renal transplantation.
3. Patients who are prevented from having blood and blood products according to a system of beliefs (e.g. Jehovah's Witnesses).
4. Patients with a pre-existing sepsis or organ injury defined as documented sepsis, acute kidney injury, acute lung injury, myocardial infarction, low cardiac output, liver injury, stroke or pancreatitis within 5 days of surgery.
5. Pregnancy.
6. Patients who are participating in another interventional clinical study.
7. Patients requiring irradiated blood.
8. Sickle cell anaemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Renal injury | baseline to 96 hours postoperatively
  measurement of serum creatinine
Myocardial injury | baseline to 72 hours postoperatively
  measurement of serum troponin

SECONDARY OUTCOMES:
Protocol compliance measured through protocol deviations | from date of randomisation through to study completion (3 months)
  protocol deviations will be aggregated based on pre-defined codes
Recruitment | from date of randomisation through to study completion (3 months)
  measured through recruitment figures
Event rates | from date of randomisation through to study completion (3 months)
  measured through serious adverse event (SAE)/ serious unexpected serious adverse reaction (SUSAR) reporting
Blinding | from date of randomisation through to study completion (3 months)
  measured through protocol deviations
Urinary neutrophil gelatinase associated lipocalin (NGAL) | baseline to 48 hours postoperatively
  measured through urine collection
Serum creatinine | at 6 weeks postoperatively
  measured to assess renal function
eGFR | at 6 weeks postoperatively
  measured to assess renal function
Sepsis-related Organ Failure Assessment (SOFA) Score | at baseline, 24, 48, 72 and 96 hours postoperatively
  Sepsis will be defined as suspected or documented infection and an acute change in total SOFA score ≥2 points consequent to the infection.
Arterial serum lactate | 24 hours postoperatively until time of resolution of hyperlactataemia
Lung injury | baseline to 96 hours postoperatively
  arterial alveolar oxygen ratios
GI tract injury | at baseline, 24, 48, 72, and 96 hours postoperatively
  serum amylase and liver function tests
Transfusion reactions | from date of randomisation through to study completion (3 months)
  measured as part of standard care to assess transfusion safety
Age of each unit of red cells transfused | day of operation
Postoperative blood loss, transfusion of red cell and non-red cell allogenic blood components | day of operation
Adverse events other than those included in the primary endpoint | from date of randomisation through to study completion (3 months)
Length of ICU and hospital stay | from date of randomisation through to study completion (3 months)

OTHER OUTCOMES:
Acute lung injury | from date of randomisation through to study completion (3 months)
  To inform the design of a subsequent efficacy trial
Acute kidney injury | from date of randomisation through to study completion (3 months)
  To inform the design of a subsequent efficacy trial
Low cardiac output | from date of randomisation through to study completion (3 months)
  To inform the design of a subsequent efficacy trial
Acute brain injury | from date of randomisation through to study completion (3 months)
  To inform the design of a subsequent efficacy trial
Acute liver or gut injury | from date of randomisation through to study completion (3 months)
  To inform the design of a subsequent efficacy trial
Sepsis | from date of randomisation through to study completion (3 months)
  To inform the design of a subsequent efficacy trial
Organ injury, sepsis or death (a composite of sepsis, acute kidney injury, acute lung injury, acute brain injury, low cardiac output syndrome, gut or liver injury or death) | from date of randomisation through to study completion (3 months)
  To inform the design of a subsequent efficacy trial
Endothelial function, tissue hypoxia and p50 of circulating red cells | baseline and 24 hours post-op
  To be measured in a sub-study of mechanisms in 80 participants
Recipient platelet, monocyte and endothelial activation in whole blood as determined using flow cytometry | baseline to 48 hours post-op
  To be measured in a sub-study of mechanisms in 80 participants
Bronchial aspirate neutrophil and protein concentration | 4-6 hours post-op
  To be measured in a sub-study of mechanisms in 80 participants
free haem | baseline to 96 hours post-op
  To be measured in a sub-study of mechanisms in 80 participants
serum bilirubin | baseline to 96 hours post-op
  To be measured in a sub-study of mechanisms in 80 participants
transferrin saturation | baseline to 96 hours post-op
  To be measured in a sub-study of mechanisms in 80 participants
non-transferrin bound iron | baseline to 96 hours post-op
  To be measured in a sub-study of mechanisms in 80 participants
hepcidin | baseline to 96 hours post-op
  To be measured in a sub-study of mechanisms in 80 participants
pulmonary leucocyte haem oxygenase-1 expression | baseline to 96 hours post-op
  To be measured in a sub-study of mechanisms in 80 participants
serum protein carbonylation and lipid peroxidation | baseline to 96 hours post-op
  To be measured in a sub-study of mechanisms in 80 participants

CONTACTS AND LOCATIONS:
Overall Officials: Gavin J Murphy, Prof, Principal Investigator — University of Leicester
Locations (1):
- Department of Cardiovascular Sciences, Leicester, Leicestershire, United Kingdom